CLINICAL TRIAL: NCT00193999
Title: Do Nasogastric Tubes After Cardiac Surgery Reduce Nausea and Vomiting. A Prospective Randomized Clinical Trial.
Brief Title: Do Nasogastric Tubes After Cardiac Surgery Reduce Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: George Djaiani, Toronto General Hospital, University Health Network
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 02-0601-B
Record Dates: First submitted 2005-09-15; First posted 2005-09-19 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2008-09

CONDITIONS: Heart Disease
Keywords: Nasogastric Tubes; Nausea; Vomiting; Cardiac surgery
MeSH Terms: conditions — Heart Diseases; Nausea; Vomiting

INTERVENTIONS:
Device: Placement of nasogastric tube

SUMMARY:
Gastric emptying is delayed after cardiac surgery, but the efficacy of the nasogastric (NG) tube in preventing distension and reducing vomiting is unclear. Nasogastric (NG) tubes are routinely used in patients undergoing surgery. They are presumed to reduce postoperative nausea and vomiting (PONV) and to lessen the risk of aspiration by reducing residual gastric volumes; however, their insertion and use is not however without potentially serious complications. Existing literature does not address their efficacy in reducing PONV after cardiac surgery. However, current evidence suggests that up to 50% of patients in this group suffer significant nausea and vomiting. The objective of this study is to determine whether NG tubes should continue to be inserted routinely during cardiac surgery to reduce PONV.

ELIGIBILITY:
Inclusion Criteria:

* undergoing coronary artery bypass graft and/or valvular surgery,
* age 18-80 year olds
* signed informed consent
* elective or urgent surgery

Exclusion Criteria:

* past history of oesophageal surgery, oesophageal varices or stricture,
* patients who have received antiemetic medication in the 24 hours before surgery
* emergency surgery
* patients that require re-sternotomy, or are not extubated 24 hours after admission to the intensive care unit, will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2003-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures will be the incidence and severity of postoperative nausea and vomiting as well as paint while the patient is in the CVICU

CONTACTS AND LOCATIONS:
Overall Officials: George Djaiani, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Djaiani G, Katznelson R, Fedorko L, Rao V, Green R, Carroll J, Katski J. Early benefit of preserved cognitive function is not sustained at one-year after cardiac surgery: a longitudinal follow-up of the randomized controlled trial. Can J Anaesth. 2012 May;59(5):449-55. doi: 10.1007/s12630-012-9675-y. PMID 22290354